CLINICAL TRIAL: NCT05799755
Title: Nintedanib Plus Standard of Care Immunosuppression Versus Standard of Care Immunosuppression Alone in Patients With Progressive Fibrotic Myositis Associated - Interstitial Lung Disease: A Randomized, Double-Blind, Exploratory Trial
Brief Title: Myositis Interstitial Lung Disease Nintedanib Trial
Acronym: MINT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rohit Aggarwal, MD (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Rohit Aggarwal, MD, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY22090061
Record Dates: First submitted 2023-02-15; First posted 2023-04-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Myositis Associated Interstitial Lund Disease (MA-ILD)
Keywords: Myositis associated interstitial lung disease (Myositis ILD); Interstitial Lung Disease (ILD); Myositis
MeSH Terms: conditions — Lung Diseases, Interstitial; Myositis | interventions — nintedanib; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 for nintedanib: placebo and stratified by underlying immunosuppressive therapy (mycophenolate vs. others). All patients must be on the standard of care (SOC) immunosuppression (IS) at screening as per the protocol and should remain on stable doses throughout the trial. After 12 weeks both arms will receive an additional 12 weeks of nintedanib (150 mg twice a day, maximum dose of 300 mg a day) through week 24 (final study visit).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators, and everyone involved in trial conduct or analysis or with any other interest in this double-blind trial will remain blinded with regard to the randomized treatment assignments until after the database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo plus Standard of Care, then Nintedanib plus Standard of Care (Placebo Comparator): Placebo twice a day (BID) plus standard of care (SOC) Immunosuppressive Therapy for 12 weeks followed by open-label Nintedanib 150 mg BID + SOC Immunosuppressive Therapy for additional 12 weeks.
  Interventions: Drug: Nintedanib; Drug: Placebo; Drug: Standard of Care
- Nintedanib plus Standard of Care (Active Comparator): Nintedanib 150 mg BID + SOC Immunosuppressive Therapy for 12 weeks followed by open-label Nintedanib 150mg BID + SOC Immunosuppressive Therapy for additional 12 weeks.
  Interventions: Drug: Nintedanib; Drug: Standard of Care

INTERVENTIONS:
Drug: Nintedanib — Nintedanib 150 mg BID
  Other Names: OFEV
Drug: Placebo — Placebo comparator
  Arms: Placebo plus Standard of Care, then Nintedanib plus Standard of Care
Drug: Standard of Care — Maximum of 2 standard of care immunosuppressant (IS) drugs are allowed, one being a glucocorticoid (GC) and the other being a non-GC IS drug OR 2 non-GC IS drugs in the event that the patient is not on a GC). The patient should be on the IS drug(s) for at least 12 weeks (at least 4 weeks or more for GC) before the screening. The doses should be stable for at least 4 weeks (at least 2 weeks for GC) before the screening visit.

SUMMARY:
This research study will evaluate safety and how well the study drug, nintedanib improve symptoms in participants with myositis associated interstitial lung disease (MA-ILD). Interstitial lung disease is a disorder caused by the abnormal accumulation of cells structures between air sacs of the lungs resulting in thickening, stiffness and scarring of the tissues of the lung.

This study will enroll a total of 134 participants across 15 clinical sites located in the United States. A subset of participants will be enrolled remotely via telemedicine utilizing certified mobile home research nurses and various remote monitoring devices.

The research visits may include a physical exam, vital signs (such as blood pressure, heart rate, etc.), pulmonary function tests (PFT and/or home spirometry), Computerized Tomography (or CT) scans of the chest, blood draws, wearing a physical activity monitor and completing questionnaires. Some of these events may be done at home, at a local facility or remotely (via telemedicine).

DETAILED DESCRIPTION:
Participants enrolled in the study will receive either study drug or placebo for 12 weeks plus the participant's normal standard of care medication for the participant's disease. Placebo is an inactive substance that contains no medicine. Following the initial treatment phase, participants will receive the active study drug (nintedanib) for an additional 12-week period.

Nintedanib is a drug that is currently used and has been approved by the Food and Drug Administration (FDA) for the treatment of idiopathic pulmonary fibrosis (IPF), and has been shown to slow the rate of decline in pulmonary function among patients with IPF as well as interstitial lung disease (ILD) associated with systemic sclerosis or scleroderma. In addition, in March 2020, the FDA approved nintedanib oral capsules to treat patients with chronic fibrosing (scarring) interstitial lung diseases (ILD) with a progressive phenotype (trait).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. Approval from local treating physician (done at pre-screening only for remote patients as well as for local site patients not actively being managed at the local site).
3. Subject lives in the United States
4. Adult: Age ≥ 18 years
5. Subject can speak, read, and understand English or Spanish
6. Subject is willing and capable of performing all study procedures.
7. Validity/repeatability of home spirometry confirmed by PFT lab technician/MD through telemedicine as per American Thoracic Society guidelines.
8. Men and women of reproductive potential must agree to use 2 reliable methods of birth control during the trial period.
9. Clinical diagnosis of myositis or presence of one of the following myositis-specific or -associated autoantibodies).

   1. Anti-synthetase autoantibody (Anti-Jo-1, -PL-7, -PL-12, -EJ, -OJ, -KS, -Tyr, -Zo)
   2. Anti-MDA5, TIF1-gamma, Mi-2, NXP2/MJ, SAE, HMGCR, SRP
   3. Anti-PM/Scl, Ku, U1RNP, Ro5,2/60, or SSA (in absence of clinical diagnosis of systemic sclerosis or primary Sjogren syndrome).
10. Fibrosing Interstitial Lung Disease (ILD):

    1. HRCT chest within 12 months of screening visit with fibrosing ILD (reticular changes, traction bronchiectasis, and/or honeycombing)
    2. No other identifiable cause of fibrosis
    3. The following co-existing features are expected and accepted: ground glass opacity, upper lung or peri-bronchovascular predominance, mosaic attenuation, air trapping, consolidation, and centrilobular nodules.
11. Progressive ILD: Defined as meeting ≥1 of the following criteria within 24 months of the screening visit.

    1. ≥10% relative decline in FVC% predicted (%pred)
    2. ≥5 but <10% relative decline in FVC %pred with worsening dyspnea.
    3. ≥5 but <10% relative decline in FVC %pred with worsening chest HRCT fibrotic changes
    4. Worsening dyspnea with worsening chest HRCT fibrosis
    5. Worsening dyspenea with FCV% </= 70%
12. Standard of care (SOC) therapy: (See: SOC immunosuppression and washout under section 6.2 for details)

    1. Allowable SOC includes a maximum of 2: 1 glucocorticoid (GC) and 1 Non-GC immunosuppressive medication (IS) Or 2 Non-GC immunosuppressive medications.
    2. Allowable IS component of SOC regimen must have been started at least 12 weeks prior and be stable for at least 4 weeks before baseline visit.
    3. In case a patient is not on any of the SOC immunosuppression, patient can be enrolled if at least 2 SOC immunosuppression are either previously failed or had intolerance or are contra-indicated.
    4. Allowable GC component of SOC regimen must have been started at least 4 weeks prior and be stable for at least 2 weeks before baseline visit.
    5. Allowable IS and GC:

       Glucocorticoid (maximum dose ≤20 mg/day; prednisone equivalent). Mycophenolate mofetil (max dose 3 gm/day) Mycophenolic acid (max dose 2,160 mg/day) Azathioprine (max dose 2.5 mg/kg/day) Methotrexate (max dose 25 mg/week Tacrolimus (max dose 10 mg/day) Cyclosporine (max dose 200 mg/day) Leflunomide (max dose 20 mg/day) Sulfasalazine (max dose 3 gm/day) JAK inhibitors (tofacitinib max does 11 mg/day, upadacitinib max dose 15 mg/day, baricitinib max does 4 mg/day) IVIG (Intravenous immunoglobulin) or SQIG (subcutaneous immunoglobulin) (max dose 2 gm/kg/month) is allowed and not considered as SOC IS therapy Rituximab (maximum dose 1000 mg x 2 (2 weeks apart) or 375mg/m2 weekly dose x 4, repeated every > 4 months) Hydroxychloroquine is allowed and not considered as SOC IS therapy. Orencia (max dose of 125 mg SQ once a week or 1 gm monthly IV infusion)
    6. Inhaled medication(s) for lung disease is allowed if started > 4 weeks before screening.

    Should remain stable throughout the study.
13. Negative pregnancy test

Exclusion Criteria:

1. Planned major surgical procedures within the trial period of 24 weeks.
2. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
3. Women of childbearing potential* not willing or able to use at least two highly effective methods of birth control.

   1. For females of reproductive potential: use of highly effective contraception for at least 1 month before study drug administration and agreement to use such a method during study participation and for an additional 28 days after the end of study drug administration.
   2. For males of reproductive potential**: use of condoms or other methods to ensure effective contraception with a partner

   Highly effective contraception examples are:
   * An approved hormonal contraceptive such as oral contraceptives, emergency contraception used as directed, patches, implants, injections, rings, hormonally-impregnated intrauterine device (IUD), or nonhormonal IUD.
   * Abstinence
   * Condoms

     * A woman is considered of childbearing potential, i.e. fertile, following menarche, and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, tubal occlusion, and bilateral oophorectomy.

       * A man is considered permanently sterile if a vasectomy has been performed.
4. Severe lung disease is defined by the following within the last 6 months before the screening:

   1. FVC ≤40 percent predicted
   2. DLCO <30% of percent predicted (corrected for Hb)
   3. O2 requirement of ≥10 L at rest based on home oxygen prescription.
   4. Patient listed for lung transplant or actively going through lung transplant evaluation.
5. Moderate to severe active muscle disease from myositis as per any one of the criteria:

   1. Creatine kinase (CK) > 2000 U/mL.
   2. Moderate to severe dermatomyositis rashes as per investigator evaluation (if rash present)
   3. Moderate to severe arthritis as per investigator evaluation
   4. Moderate to severe muscle weakness as per Sit to Stand 30 seconds of < 7.
6. History of or ongoing serious active, chronic, or recurrent infection within 4 weeks of screening
7. Significant Pulmonary Hypertension (PH) is defined by any of the following:

   1. Current clinical diagnosis of moderate to severe PH or significant right heart failure.
   2. History of echocardiographic evidence of significant right heart failure or moderate to severe PH (TR jet >= 2.9 m/s and signs of right ventricle (RV) dysfunction; or TR jet > 3.4; or an right ventricle systolic pressure (RVSP) > 40-55 with evidence of RV strain or dysfunction; or RVSP > 55 regardless.
   3. History of right heart catheterization showing a cardiac index ≤ 2.2 l/min/m² or severity of pulmonary hypertension (mPAP) >40 millimeters of mercury (mmHg) with a pulmonary capillary wedge pressure (PCWP) <15mmHg
   4. PH requiring oral, IV, or inhaled therapy (such as epoprostenol, treprostinil, iloprost, bosentan, ambrisentan, sildenafil, and tadalafil).
8. Increased bleeding risk, defined by any of the following:

   1. Patients who require

      * Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, factor Xa inhibitors, low molecular weight heparin)
      * High dose antiplatelet therapy (>325mg acetylsalicylic acid or >75mg clopidogrel).
   2. History of hemorrhagic central nervous system (CNS) event within 12 months of screening.
   3. Any of the following within 3 months of screening:

      * Hemoptysis or hematuria
      * Active gastrointestinal (GI) bleeding or active GI ulcers.
   4. Coagulation parameters: International normalized ratio (INR) >2, prolongation of prothrombin time (PT) and by >1.5 x ULN at screening.
9. History of a thrombotic event (including stroke and transient ischemic attack) within 12 months of screening.
10. Severe Cardiovascular disease, any of the following:

    1. Severe hypertension, uncontrolled under treatment (≥160/100 mmHg), within 6 months of screening.
    2. Myocardial infarction or unstable cardiac angina within 6 months of screening.
11. Patients with underlying chronic liver disease (Child-Pugh A, B, or C hepatic impairment).
12. Known hypersensitivity to the trial medication or its components (i.e. soya lecithin)
13. Other diseases that may interfere with testing procedures or in the judgment of the Investigator may interfere with trial participation (such as significant GI issues like irritable bowel syndrome, inflammatory bowel disease, recent abdominal surgery, diverticular disease), or significant other lung diseases (such as severe obstructive lung disease such as severe asthma or severe chronic obstructive pulmonary disease, etc.) or may put the patient at risk when participating in this trial.
14. Life expectancy for a disease other than ILD < 2.5 years (Investigator assessment).
15. In the opinion of the investigator, any condition precluding participation and completion of the study, including active alcohol and drug abuse or patients not able to understand or follow trial procedures.
16. Other investigational therapy was received within 1 month or 6 half-lives (whichever was greater) before the screening visit.
17. Current treatment with nintedanib or pirfenidone (taken the drug within 3 months of randomization or history of intolerance/side effects)
18. Current or recent use of one or more of the following medications (See: SOC immunosuppression and washout under section 6.2 for details)

    1. Cyclophosphamide within 3 months of baseline.
    2. Anti-tumor necrosis factor (infliximab, golimumab, or certolizumab) within 8 weeks or adalimumab within 4 weeks, and etanercept within 2 weeks of baseline.
    3. Anakinra within 1 week of baseline.
    4. Other biological agents such as tocilizumab, etc. within 4 weeks of baseline.
19. Safety laboratory abnormality as any one of below

    1. Aspartate transferase (AST), alanine aminotransferase (ALT) > 1.5 x ULN at screening, unless deemed due to active myositis by investigator, in which case CK is also abnormally elevated and the ratio of AST or ALT by CK levels (adjusted as x ULN) should be < 2.0 and gamma-glutamyl transferase < 2.0 x ULN.
    2. Bilirubin > 1.5 x ULN at screening
    3. Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula at screening.
    4. Hgb < 9.0
    5. Platelet count < 100,000/mm3
    6. White blood cells < 3000/mm3

       -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (L-PF) Dyspnea score | Baseline (week 0) to 12 weeks
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules: Symptoms (23 items) and Impacts (21 items).
  The Symptoms module yields three domain scores: 1) dyspnea, 2) cough and 3) fatigue as well as a total Symptoms score. The Impacts module yields a single Impacts score. Symptoms and Impacts scores are summed to yield a total L-PF score. Scoring is performed as a summary score, the mean of the dimension ratings multiplied by 100. Summary score range from 0-100, the higher the score the greater the impairment.

SECONDARY OUTCOMES:
Change in Living with Pulmonary Fibrosis Dyspnea score | Baseline (week 0) to week 24
  The Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules: Symptoms (23 items) and Impacts (21 items).
  The Symptoms module yields three domain scores: 1) dyspnea, 2) cough and 3) fatigue as well as a total Symptoms score. The Impacts module yields a single Impacts score. Symptoms and Impacts scores are summed to yield a total L-PF score. Scoring is performed as a summary score, the mean of the dimension ratings multiplied by 100. Summary score range from 0-100, the higher the score the greater the impairment.
Change in other Living with Pulmonary Fibrosis scores | Week 12 to week 24
  The Living with Pulmonary Fibrosis questionnaire (L-PF) scores will include total score, symptoms, cough, energy and impacts scores. The score range is from 0-100, the higher the score, the greater the impairment.
Change in immunosuppressive (IS) regimen | Baseline (Week 0) to week 12
  Proportion of patients requiring an increased dose or a change in their glucocorticoid (GC) / immunosuppression (IS) agent for clinical worsening/flare of MA-ILD
Absolute and relative change in Forced Vital Capacity (FVC) (mL) from baseline to 12 weeks | Baseline (week 0) to week 12
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml.
Absolute and relative change in Forced Vital Capacity (FVC) (mL) from baseline to 24 weeks | Baseline (week 0) to week 24
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml.
Absolute and relative change in Forced Vital Capacity FVC (%) from baseline to week 12 | Baseline (week 0) to week 12
  FVC (%) is forced vital capacity parameter derived from a pulmonary function study (PFT)as percentage predicted of healthy standards (in %), respectively.
Absolute and relative change in Forced Vital Capacity FVC (%) from baseline to week 24 | Baseline (week 0) to week 24
  FVC (%) is forced vital capacity parameter derived from a pulmonary function study (PFT)as percentage predicted of healthy standards (in %), respectively.
Proportion of patients with a relative decline from baseline in FVC (mL) of ≥10%, ≥7.5%, and ≥ 5% | Weeks 12 and 24
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively.
Proportion of patients with stable (+/- < 5%) or improved FVC (≥ 5, ≥ 7.5, ≥ 10%) (mL) from baseline to week 12 | baseline (week 0) at week 12
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Percent change is calculated based on change from baseline to a follow up visit.
Proportion of patients with stable (+/- < 5%) or improved FVC (≥ 5, ≥ 7.5, ≥ 10%) (mL) from baseline to week 24 | baseline (week 0) at week 24
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Percent change is calculated based on change from baseline to a follow up visit.
Time to FVC (mL) improvement and decline from baseline by (≥5%, 7.5%, 10%) | Baseline (week 0) to 24 weeks
  FVC (ml) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Time to designated change is calculated based on change from baseline to a follow up visit and time since baseline.
Time to progression | Baseline (week 0) to week 24
  Defined as either time for event a, b or c Event a. ≥ 10% decline in FVC (mL) or death or transplant Event b. ILD worsening definition (per protocol) or death or transplant Event c. non-elective hospitalization for ILD worsening/flare or death or lung transplant
Proportion of patients with stable (+/- < 5%) or improved FVC (≥ 5, ≥ 7.5, ≥ 10%) (%) from baseline to week 12 | baseline (week 0) at week 12
  FVC (%) are forced vital capacity parameter derived from a pulmonary
Proportion of patients with stable (+/- < 5%) or improved FVC (≥ 5, ≥ 7.5, ≥ 10%) (%) from baseline to week 24 | baseline (week 0) at week 24
  FVC (%) are forced vital capacity parameter derived from a pulmonary
Proportion of patients with a relative decline from baseline in FVC (%) of ≥10%, ≥7.5%, and ≥ 5% | Weeks 12 and 24
  FVC (%) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively.
Time to FVC (%) improvement and decline from baseline by (≥5%, 7.5%, 10%) | Baseline (week 0) to 24 weeks
  FVC (%) is forced vital capacity parameter derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Time to designated change is calculated based on change from baseline to a follow up visit and time since baseline.

OTHER OUTCOMES:
Rate of patient recruitment, enrollment, screen failure, and dropout rates between the local sites (average per site) and the remote site | Baseline (week 0) to week 24
  Compare the patient recruitment, enrollment, screen failure and drop out rates between patient recruited through local clinical trial sites vs. remote clinical trial site.
Reliability measure of Forced Vital Capacity (FVC) in ml measured by home spirometry | Baseline (week 0) to week 24
  Reliability is measured as test (baseline) and re-test (week 1) correlation of FVC in ml using spearman correlation.
Validity of Forced Vital Capacity (FVC) in ml by home spirometry | Baseline (week 0) to week 24
  Validity of FVC (ml) by home spirometry is measured as spearman correlation with FVC (ml) obtained by gold standard clinic spirometry.
Absolute and relative change in DLCO | Baseline (week 0) to week 24
  DLCO is diffusing capacity of the lungs for carbon monoxide (DLCO) derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Changes from baseline to follow up will be calculated and compared between two treatment arms.
Progression free survival | weeks 12 and 24
  Connective Tissue Disease (CTD)-ILD outcome as per Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT), which is defined as the occurrence of any of the following: death or lung transplant or FVC ≥10% decline or FVC ≥5% decline with DLCO ≥15% decline Clinical worsening is defined as death, lung transplant, or new/worsening O2 requirement at rest (>2L), or non-elective hospitalization for ILD clinical worsening/flare or ILD worsening definition (per protocol) or out of protocol rescue medication for ILD clinical worsening/flare.
Steroid use (calculated using prednisone dose equivalents) | Weeks 12 and 24
  Comparing change of steroid from baseline to follow up, between 2 treatment groups
Change in supplemental oxygen needs from baseline to week 12 | Baseline (week 0) to 12 weeks
  Comparing change in oxygen requirement from baseline to follow up, between 2 treatment groups
Mean change in supplemental oxygen requirement in ml from baseline to week 24 | Baseline (week 0) to 24 weeks
  Comparing change in oxygen requirement from baseline to follow up, between 2 treatment groups
Patient assessment of change | Weeks 12 and 24
  Patient Assessment of Change (also known as Patient Global Impression of Change): Overall Assessment of Change by Patient. Patient overall assessment of change in disease status from baseline, reported as 7-point ordinal scale: no change, minimal, moderate, and major worsening as well as minimal, moderate and major improvement.
Physician assessment of change | Weeks 12 and 24
  Physician's overall assessment of change in disease status of the patient from baseline, reported as 7-point ordinal scale: no change, minimal, moderate, and major worsening as well as minimal, moderate and major improvement.
Change in Cadence by Physical Activity Monitor at week 12. | Baseline (week 0) to 12 weeks
  Cadence: highest step counts performed in a minute for a given day. Higher value is better.
  Mean change in cadence from baseline to week 12.
Change in Average Daily Step Count by Physical Activity Monitor at week 12. | Baseline (week 0) to 12 weeks
  Average daily step count measured by mean of daily step count for 7 days, where daily step counts in a day divided by time the device was worn. Higher value is better.
  Mean change in average daily step count from baseline to week 12
Change in Cadence by Physical Activity Monitor at week 24. | Baseline (week 0) to 24 weeks
  Cadence: highest step counts performed in a minute for a given day. Higher value is better.
  Mean change in cadence from baseline to week 24.
Change in Average Daily Step Count by Physical Activity Monitor at week 24. | Baseline (week 0) to 24 weeks
  Average daily step count measured by mean of daily step count for 7 days, where daily step counts in a day divided by time the device was worn. Higher value is better.
  Mean change in average daily step count from baseline to week 24.
Changes in Sit to Stand test from baseline to week 12 | Baseline (week 0) to 12 weeks
  Evaluate the changes in Sit to Stand test score from baseline to follow up , between two treatment arms
Changes in Sit to Stand test from baseline to week 24 | Baseline (week 0) to 24 weeks
  Evaluate the changes in Sit to Stand test score from baseline to follow up , between two treatment arms
Change in High-Resolution Computed Tomography (HRCT) chest from baseline | Baseline (week 0) to 24 weeks
  Change in HRCT will be analyzed using semi-quantitative and quantitative image based scoring. Change from baseline to follow up will be calculated and compared between two treatment arm
Adverse events (AEs) and tolerance | Baseline (week 0) to week 24
  All AEs and tolerance event will be compared between 2 treatment arms
  * Proportion of subjects who discontinue study drug
  * Patients with any AEs
  * Patients with Serious Adverse Event (SAE)s
  * Patients with AEs of special interest (gastrointestinal perforation and hepatic injury)
Absolute and relative change in FEV1 | Baseline (week 0) to week 24
  FEV1 is forced expiratory volume over 1 second (FEV1) derived from a pulmonary function study (PFT) in volume as ml and as percentage predicted of healthy standards (in %), respectively. Changes from baseline to follow up will be calculated and compared between two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Aggarwal, MD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - National Jewish Health, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Columbia University Irving Medical Center, New York, New York
  - Northwell Health, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Sharing of individual participant data will require written approval from sponsor and steering committee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests will not be accepted prior to final publication of the trial.
Access Criteria: All data requests will require written approval from sponsor and steering committee prior to release of data

REFERENCES:
- [Background] Distler O, Highland KB, Gahlemann M, Azuma A, Fischer A, Mayes MD, Raghu G, Sauter W, Girard M, Alves M, Clerisme-Beaty E, Stowasser S, Tetzlaff K, Kuwana M, Maher TM; SENSCIS Trial Investigators. Nintedanib for Systemic Sclerosis-Associated Interstitial Lung Disease. N Engl J Med. 2019 Jun 27;380(26):2518-2528. doi: 10.1056/NEJMoa1903076. Epub 2019 May 20. PMID 31112379
- [Background] Flaherty KR, Wells AU, Cottin V, Devaraj A, Walsh SLF, Inoue Y, Richeldi L, Kolb M, Tetzlaff K, Stowasser S, Coeck C, Clerisme-Beaty E, Rosenstock B, Quaresma M, Haeufel T, Goeldner RG, Schlenker-Herceg R, Brown KK; INBUILD Trial Investigators. Nintedanib in Progressive Fibrosing Interstitial Lung Diseases. N Engl J Med. 2019 Oct 31;381(18):1718-1727. doi: 10.1056/NEJMoa1908681. Epub 2019 Sep 29. PMID 31566307
- [Background] Wilfong EM, Aggarwal R. Role of antifibrotics in the management of idiopathic inflammatory myopathy associated interstitial lung disease. Ther Adv Musculoskelet Dis. 2021 Dec 9;13:1759720X211060907. doi: 10.1177/1759720X211060907. eCollection 2021. PMID 34917177
- [Background] Shen L, Yan Q, Chen X. Efficacy of Combination Therapy With Pirfenidone and Low-Dose Cyclophosphamide for Refractory Interstitial Lung Disease Associated With Connective Tissue Disease: A Case-Series of Seven Patients. Arch Rheumatol. 2019 Aug 26;35(2):180-188. doi: 10.46497/ArchRheumatol.2020.7381. eCollection 2020 Jun. PMID 32851366
- [Background] Li T, Guo L, Chen Z, Gu L, Sun F, Tan X, Chen S, Wang X, Ye S. Pirfenidone in patients with rapidly progressive interstitial lung disease associated with clinically amyopathic dermatomyositis. Sci Rep. 2016 Sep 12;6:33226. doi: 10.1038/srep33226. PMID 27615411
- [Background] Khanna D, Mittoo S, Aggarwal R, Proudman SM, Dalbeth N, Matteson EL, Brown K, Flaherty K, Wells AU, Seibold JR, Strand V. Connective Tissue Disease-associated Interstitial Lung Diseases (CTD-ILD) - Report from OMERACT CTD-ILD Working Group. J Rheumatol. 2015 Nov;42(11):2168-71. doi: 10.3899/jrheum.141182. Epub 2015 Mar 1. PMID 25729034
- [Background] Liang J, Cao H, Yang Y, Ke Y, Yu Y, Sun C, Yue L, Lin J. Efficacy and Tolerability of Nintedanib in Idiopathic-Inflammatory-Myopathy-Related Interstitial Lung Disease: A Pilot Study. Front Med (Lausanne). 2021 Feb 3;8:626953. doi: 10.3389/fmed.2021.626953. eCollection 2021. PMID 33614683
- [Derived] Aggarwal R, Oddis CV, Sullivan DI, Moghadam-Kia S, Saygin D, Kass DJ, Koontz DC, Li P, Conoscenti CS, Olson AL; MINT investigators. Design of a randomised controlled hybrid trial of nintedanib in patients with progressive myositis-associated interstitial lung disease. BMC Pulm Med. 2024 Oct 30;24(1):544. doi: 10.1186/s12890-024-03314-0. PMID 39478532